CLINICAL TRIAL: NCT01228578
Title: Multi-vitamins, HAART and HIV/AIDS in Uganda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Makerere University (Other); Infectious Disease Institute, Kampala, Uganda (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD060333-01
Record Dates: First submitted 2010-10-15; First posted 2010-10-26 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: HIV/AIDS
Keywords: Multivitamins; HIV/AIDS; Immune reconstitution; Weight Gain; Quality of Life
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Weight Gain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multivitamins (B,C,E) (Experimental)
  Interventions: Dietary Supplement: Multivitamin supplements B,C and E
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Multivitamin supplements B,C and E

INTERVENTIONS:
Dietary Supplement: Multivitamin supplements B,C and E — One daily recommended dietary allowance of multivitamins B,C and E or placebo taken daily for 18 months

SUMMARY:
The investigators are conducting a double-blind, placebo controlled,randomized trial of multivitamin supplements(containing B-vitamins, C, and E) to determine their efficacy in slowing disease progression, indicated by increased CD4 count, weight gain, and improved quality of life, and decreased morbidity, mortality, and drug-related adverse events (i.e. peripheral neuropathy, anemia, and diarrhea).

The investigators hypothesize that daily multivitamin supplementation will: (1) improve immune reconstitution; (2) improve weight gain, and (3) improve quality of life.

DETAILED DESCRIPTION:
Antiretroviral therapy, gradually becoming the standard of care in developing countries, confers enormous benefits and yet substantial morbidity remains in human immunodeficiency virus (HIV) positive populations. Multivitamin supplements have immune-enhancing effects, and supplements were found to improve immunologic status and reduce morbidity and mortality among HIV-positive Tanzanian women in pre-highly active anti-retroviral therapy (HAART) stages of disease. These supplements are thought to be required to restore adequate nutrient levels in the context of HIV infection.

This study will enroll 400 men and women in the Kampala district of Uganda, who are receiving or have recently initiated HAART. At baseline and monthly thereafter, research physicians and nurses at study clinics will assess each participant's clinical status and undertake study procedures. Each participant will be followed for 18 months, or until his/her death or loss to follow-up. Home visits will be conducted if participants miss their scheduled clinic appointments. We will perform nutritional assessments (anthropometry and dietary intake) at enrollment and several follow-up points, and laboratory measurements (CD4 cell counts and complete blood counts) every six months.

Importantly, all study participants will continue receiving the standard of care according to national guidelines for the entire study period. Multivitamins could be a low-cost, adjunct therapy for helping to alleviate disease burden and elevate quality of life in HIV-infected individuals on HAART. At the same time, their efficacy could help preserve limited drug regimens in developing settings by postponing the need for switches to second line regimens of HAART.

Our proposal represents a collaboration between the Harvard School of Public Health, Infectious Disease Institute and Makerere University School of Public Health in Kampala, Uganda.

ELIGIBILITY:
Inclusion Criteria:

* men or women aged >=18 years old
* HIV-positive
* initiating anti-retroviral therapy at the time of randomization or have been on highly active anti-retroviral therapy (HAART) for no more than 6 months
* have no intention of migrating, or re-locating >= 20 km outside of the Infectious Disease Institute (IDI), or Kiswa Health Center within the next 18 months after enrollment
* agree to allow home visit(s) and subsequent follow-up contacts as part of the study
* provide written informed consent

Exclusion Criteria:

* pregnant Women
* individuals from whom we are unable to obtain written informed consent will be excluded from the study. For example, patients that are extremely ill and unable to consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Weight Gain | 18 months
Immune Reconstitution | 18 months
  Immune Reconstitution is measured by change in CD4 cell count
Improved Quality of Life | 18 months

SECONDARY OUTCOMES:
New or recurrent disease progression event | 18 months
Reduce the probability of changing drug therapy (indicated by switching from first- to second-line therapy) | 18 months
Reduce HAART-associated adverse events (indicated by incident peripheral neuropathy, severe anemia, or diarrhea). | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MD,MPH,DrPH, Principal Investigator — Harvard School of Public Health (HSPH); David Guwatudde, MPH, PhD, Principal Investigator — Makerere University
Locations (1):
- Makerere University School of Public Health / Infectious Disease Institute, Kampala, Uganda

REFERENCES:
- [Derived] Guwatudde D, Wang M, Ezeamama AE, Bagenda D, Kyeyune R, Wamani H, Manabe YC, Fawzi WW. The effect of standard dose multivitamin supplementation on disease progression in HIV-infected adults initiating HAART: a randomized double blind placebo-controlled trial in Uganda. BMC Infect Dis. 2015 Aug 19;15:348. doi: 10.1186/s12879-015-1082-x. PMID 26285704
- [Derived] Guwatudde D, Ezeamama AE, Bagenda D, Kyeyune R, Wabwire-Mangen F, Wamani H, Mugusi F, Spiegelman D, Wang M, Manabe YC, Fawzi WW. Multivitamin supplementation in HIV infected adults initiating antiretroviral therapy in Uganda: the protocol for a randomized double blinded placebo controlled efficacy trial. BMC Infect Dis. 2012 Nov 15;12:304. doi: 10.1186/1471-2334-12-304. PMID 23151221